CLINICAL TRIAL: NCT03529201
Title: Effectiveness of Quadratus Lumborum Block After Nephrectomy
Brief Title: QLB After Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Collaborators: Department of Anesthesiology and Intensive Care, F. Chopin Hospital in Rzeszów (Unknown); Department of Anesthesiology and Intensive Care, J. Śniadecki Hospital in Białystok (Unknown)
Responsible Party: Principal Investigator, Michał Borys, M.D., Ph.D., Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-0254/328/2017
Record Dates: First submitted 2018-05-01; First posted 2018-05-18 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative; Chronic Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Passive Cutaneous Anaphylaxis; Oxycodone; Sevoflurane; Fentanyl; Rocuronium

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to one of the study arms: QLB or control group.
Who Masked: Participant
Masking Description: A regional block will be performed under general anesthesia. Patients will not be aware of this procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QLB (Experimental): At the end of surgery, QLB with ropivacaine will be done on the side of the operation.
  Interventions: Procedure: QLB; Device: PCA; Procedure: GA; Drug: Oxycodone; Drug: Sevoflurane; Drug: Fentanyl; Drug: Rocuronium
- Control (Experimental): Standard care. No regional blocks.
  Interventions: Device: PCA; Procedure: GA; Drug: Oxycodone; Drug: Sevoflurane; Drug: Fentanyl; Drug: Rocuronium

INTERVENTIONS:
Procedure: QLB — On the side of the surgery, QLB with 0.375% ropivacaine (0.2 mL/kg)
  Arms: QLB
Device: PCA — Patient-controlled analgesia
Procedure: GA — General anesthesia
Drug: Oxycodone — administered by PCA
Drug: Sevoflurane — Inhalational anesthetic during GA
Drug: Fentanyl — painkiller during GA
Drug: Rocuronium — muscle relaxant during GA

SUMMARY:
Oxycodone consumption and postoperative pain intensity in patients undergoing nephrectomy procedures. Of all study participants, 50% will obtain quadratus lumborum block (QLB).

DETAILED DESCRIPTION:
Patients undergoing nephrectomy procedures will be allocated to one of the study arms. At the end of an operation, still under general anesthesia, 50% patients will obtain QLB with ropivacaine.

Ultrasound-guided QLB will be performed on the side of surgery with 0.375% ropivacaine solution (0.2 mL per kg).

Every patient will get patient-controlled analgesia pump with oxycodone in the postoperative period.

Postoperative pain will be measured with VAS (visual-analogue scale) 2, 4, 8, 12 and 24 hours after the end of the operation. 24 -hours period.

At the 1, 3, 6 months patients will be interviewed by phone to assess neuropathic pain. Neuropathic Pain Symptom Inventory (NPSI) will be used.

ELIGIBILITY:
Inclusion Criteria:

* obtained consent
* nephrectomy procedure

Exclusion Criteria:

* coagulopathy allergy to local anesthetics depression, antidepressant drugs treatment epilepsy usage of painkiller before surgery addiction to alcohol or recreational drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
Total consumption of oxycodone | 24 hours after the end of surgery.
  Overall use of oxycodone administered by PCA pump will be assessed.

SECONDARY OUTCOMES:
Pain intensity | 24 hours after the end of surgery
  Pain intensity measured on VAS scale at the 2, 4, 8, 12, 24 hours. VAS in milimmeters. Minimum value 0, maximum 100. Less better - less severe pain. 0 no pain at all.
Chronic pain | 6 months after the surgery
  Chronic pain occurrence assessed with Neuropathic Pain Symptom Inventory (NPSI) 10 descriptive variables, each one from 0 to 10. 0 means no pain. 10 very high chance of occurrence of neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Department of Anesthesiology and Intensive Care, J. Śniadecki Hospital in Białystok, Bialystok
  - Department of Anesthesiology and Intensive Care, F. Chopin Hospital in Rzeszów, Rzeszów

IPD SHARING:
Plan to Share IPD: No